CLINICAL TRIAL: NCT05841355
Title: MADRE (Mammograms Available Due to Research and Education)
Acronym: MADRE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Yamile Molina, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2022-0531
Record Dates: First submitted 2023-04-23; First posted 2023-05-03 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Screening
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Compare intervention effects on BC screening among 400 non-adherent individuals in a 1:1 empower/educate ratio (n=200 per group)
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Educate (Education + Navigation) Sessions (Other): Session 1 BC knowledge, BC disparities, USPSTF guidelines, barriers and preferred solutions to BC screening, Community Health Workers (CHW) testimonials, empirical data, individual action plans for BC screening Session 2 &3 Health knowledge (diet and physical activity guidelines), barriers and preferred solutions to dietary and physical activity change, CHW testimonials, empirical data, individual action plans for diet
  Interventions: Other: Educate
- Empower (Empowerment + Navigation) Sessions (Other): Session 1 BC knowledge, BC disparities, USPSTF guidelines, barriers and preferred solutions to BC screening CHW testimonials, Empirical data, Individual action plans for BC screening Sessions 2 & 3 BC screening as leading by example, BC promotion strategies that reflect personal and network members' preferences, opportunities to volunteer/be a part of tight-knit initiatives, partnerships with navigators/CHWs to serve as "bridges" for network members CHW testimonials , resource guides for BC promotion, individual action plans for promoting BC, role playing activities (session 2) Participant testimonials, participant relays empirical data, group discussion and plans for promoting BC (session 3)
  Interventions: Other: Empower

INTERVENTIONS:
Other: Educate — Education sessions
  Arms: Educate (Education + Navigation) Sessions
Other: Empower — Empowerment sessions
  Arms: Empower (Empowerment + Navigation) Sessions

SUMMARY:
The design builds on past studies by integrating social network analysis (SNA) and implementation science (IS) into a longitudinal randomized clinical trial (RCT). The investigator will compare the long-term effects of interventions by examining guideline-concordant initial and repeat Breast Cancer (BC) screening.

DETAILED DESCRIPTION:
To further test the added benefits of the empower approach relative to traditional educate approaches. Past community research has primarily focused on one-time BC screening among intervention participants. The design builds on past studies by integrating social network analysis (SNA) and implementation science (IS) into a longitudinal randomized clinical trial (RCT). The investigator will compare the long-term effects of interventions by examining guideline-concordant initial and repeat BC screening. The investigator will estimate the widespread effects of interventions by prospectively collecting data from network members not involved in the RCT. The investigator will also explore "active ingredients" that underlie intervention effects, including psychosocial, IS and network mechanisms. Overall, the investigator will demonstrate whether and how non-adherent individuals may "boost" intervention effects throughout their networks.

The investigator's goal is to further test the added benefits of the empower approach relative to traditional educate approaches. Past community research has primarily focused on one-time BC screening among intervention participants. The investigator's novel design builds on past studies by integrating social network analysis (SNA) and implementation science (IS) into a longitudinal randomized clinical trial (RCT). The investigator will compare the long-term effects of interventions by examining guideline-concordant initial and repeat BC screening. The investigator will estimate the widespread effects of interventions by prospectively collecting data from network members not involved in the RCT. The investigator will also explore "active ingredients" that underlie intervention effects, including psychosocial, IS and network mechanisms. Overall, the investigator will demonstrate whether and how non-adherent individuals may "boost" intervention effects throughout their networks.

Aim 1: Among 400 non-adherent individuals, the investigator will compare intervention effects on BC screening, using an individual RCT in a federally qualified health center (FQHC). The investigator will use the US Preventative Services Task Force (USPSTF) guidelines - i.e., 40-74 year-olds should obtain mammograms every 2 years.

Aim 2: Among 200 network members, the investigator will compare intervention effects on BC screening, based on the USPSTF guidelines.

Aim 3: The investigator will explore mechanisms of change underlying intervention effects on BC screening using IS measures, descriptive SNA, and structural equation models. If study arms are comparable, the investigator will examine which mechanisms may predict multilevel intervention effects across approaches.

ELIGIBILITY:
Aim 1

Inclusion Criteria:

* female biological sex
* identification as Latinas
* non-adherence to USPSTF guidelines (42-74 years old, no mammogram in past 2 years, no previous BC diagnosis)
* no previous history of health volunteerism
* not a network member enrolled in Aim 2.

Exclusion Criteria

* Not meeting at least one of the aforementioned Aim 1 inclusion criteria.

Aim 2.

Inclusion Criteria:

* female biological sex
* eligibility to obtain BC screenings by USPSTF guidelines (i.e., 40-74 years old, no personal BC history)
* referral from Aim 1 participants
* no previous history of health volunteerism
* no participation in the RCT (not an Aim 1 participant, no Session #3 attendance).

Exclusion Criteria:

* Not meeting at least one of the aforementioned Aim 1 inclusion criteria.

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 600 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Breast Cancer (BC) Screening (Aim 1) | 1-4 years
  Compare the number of participants in the empowerment arm that obtain guideline-concordant initial and repeat BC screening with the the number of participants in the education arm
Breast Cancer Screening (Aim 2) | 1-4 years
  Compare the number of network members in the empowerment arm that obtain guideline-concordant initial and repeat BC screening with the number of non-adherent network members in the education arm

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mile Square Health Center, Chicago, Illinois
  - University of Illinois Health, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be shared, based on correspondence between researchers. There will need to be safeguards in place to ensure privacy and confidentiality, given the nature of social network data.

REFERENCES:
- [Derived] McClellan SP, De La Paz E, Arroyo J, Montoya S, Perez J, Wright E, Moreno E, Padilla M, Kroenke CH, Rauscher GH, Neuschler E, Ganschow P, Stackhouse N, Atkins M, Dziak JJ, Neal JW, Lucio A, Molina Y. The "Mammograms Available Due to Resources and Education" (MADRE) Study: Rationale and Design. Contemp Clin Trials. 2025 Feb;149:107786. doi: 10.1016/j.cct.2024.107786. Epub 2024 Dec 22. PMID 39719248